CLINICAL TRIAL: NCT04176744
Title: Optimization of Non-invasive Diaphragm Activation Using Magnetic Phrenic Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPTISTIM_2019
Record Dates: First submitted 2019-11-19; First posted 2019-11-25 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2019-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Each participant enrolled in the study will be tested with different stimulation settings on three different days in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic Phrenic Nerve Stimulation (Experimental): Each participant will be tested with 4 different stimulation setups (coils and stimulator) on 3 different days.
  Interventions: Other: Uni- and bilateral magnetic phrenic nerve stimulation

INTERVENTIONS:
Other: Uni- and bilateral magnetic phrenic nerve stimulation — Uni- and bilateral magnetic phrenic nerve stimulation using different coils, stimulation patterns (frequency, intensity, number of pulses) and locations (neck, chest).

SUMMARY:
The use of mechanical ventilation (MV) to replace spontaneous breathing has been associated with respiratory muscle dysfunction and lung injury from positive pressure. While using MV in an intensive care unit setting, the diaphragm is unloaded, potentially resulting in early development of diaphragmatic atrophy in as early as 18 hours of complete diaphragm inactivity. These changes in muscle properties result in a decrease in the force generating capability of the muscle, ultimately resulting in difficulty to restore spontaneous breathing and a subsequent prolonged weaning process or failure. A prolonged weaning period is associated with longer duration of MV, which may result in a cascade of further diaphragm dysfunction, weakness, and injury.

Stimulation of the phrenic nerves to produce diaphragm contraction and activity is a possible mechanism to reduce MV related diaphragm dysfunction. Two promising studies have shown the potential of repetitive phrenic nerve stimulation on inducing diaphragm activity in human subjects with trains of pulses via both cervical and bilateral phrenic nerve stimulation. However, neither study provided optimal stimulation settings. As such, the primary purpose of this study is to investigate the optimal settings for noninvasive phrenic nerve stimulation to induce diaphragm contraction.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age: 18 - 35 years
* Non-smoking
* Healthy
* Able to communicate in English
* Normal lung function
* Normal Body mass index between 18.5 and 24.9 kg/m2
* Willingness to adhere to the study rules

Exclusion Criteria:

* Acute illness or chronic conditions affecting sleep or the performance of the respiratory, cardiovascular, neuromuscular, gastrointestinal or muscle system
* Women who are pregnant or breast feeding or have the intention to become pregnant during the course of the study
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Known or suspected non-compliance, drug or alcohol abuse
* Intake of medication affecting sleep or the performance of the respiratory, cardiovascular or neuromuscular system or gastrointestinal or muscle system
* Presence of cardiac pacemaker, implanted defibrillators or implanted neurostimulators
* Any metal or electronics inside of the body
* History of seizures or epilepsy
* Tattoos on the stimulation sites
* Previous enrolment into the current study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in airflow | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Flow will be recorded by a pneumotachometer and averaged over breaths.
Changes in costal diaphragm activity | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Costal diaphragm activity will be continuously recorded via a wireless surface electromyography system.
Changes in transdiaphragmatic pressure | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Transdiaphragmatic pressure changes, i.e. changes in esophageal and gastric pressures, will be measured by a pressure transducer connected to balloon-catheters.
Changes in mouth pressure | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Mouth pressure will be continuously recorded using a differential pressure transducer.
Changes in abdominal movements | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Abdominal movements will be assessed using the respiratory belt strain transducer.

SECONDARY OUTCOMES:
Changes in extradiaphragmatic muscle activity | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Muscle activity will be continuously recorded via a wireless surface electromyography system.
Changes in head, shoulder and arm movements | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Head, shoulder and arm movements will be recorded using wireless acceleration sensors.
Changes in stress related parameters (heart rate, blood pressure, skin conductance) | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Heart rate will will be continuously recorded with electrodes. Blood pressure will be continuously recorded using a non-invasive device. Skin conductance will be continuously recorded with electrodes worn on two fingers.
Perception of pain, paresthesia and distress | Assessed 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Participant subject perception of pain, paresthesia and distress will be evaluated with a visual analogue scales.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M. Spengler, Prof., Principal Investigator — Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyle KGPJM, Eichenberger PA, Schon P, Spengler CM. Inspiratory response and side-effects to rapid bilateral magnetic phrenic nerve stimulation using differently shaped coils: implications for stimulation-assisted mechanical ventilation. Respir Res. 2022 Dec 17;23(1):357. doi: 10.1186/s12931-022-02251-y. PMID 36528761